CLINICAL TRIAL: NCT02280707
Title: Grab a Cup, Fill it up! An Intervention to Promote Convenience of Drinking Water and Increase Student Water Consumption During School Lunch.
Brief Title: Intervention to Promote Water Consumption in School Lunchrooms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Catherine Giles, Project Manager, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19475-105
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Water Consumption; Schools

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Grab a Cup, Fill it Up
- Control (No Intervention)

INTERVENTIONS:
Other: Grab a Cup, Fill it Up — The intervention involved installing promotional posters encouraging students to drink water as well as cup dispensers stocked with disposable 5 ounce cups near water fountains in school lunchrooms.
  Arms: Intervention

SUMMARY:
This study, randomized, delivered, and analyzed at the school level, evaluated the effect of simple, structural changes to school lunch rooms to make drinking water easier for students during lunch time. Half of the schools received posters promoting drinking water and installed cup dispensers stocked with cups next to lunchroom water fountains, while the other half received no intervention. The intervention outcomes were average water consumption and the proportion of students in the lunchroom who opted to drink water, as well as the proportion of students with sugary drinks at lunch. No identifying information on individual children was collected.

ELIGIBILITY:
Inclusion Criteria: School in Boston Public School district in Boston, MA; had to have plumbed drinking water access in school cafeteria -

Exclusion Criteria: School had no plumbed drinking water access in cafeteria.

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in average student water consumption at lunch | March 2013-June 2013, up to 4 months

SECONDARY OUTCOMES:
Change in proportion of students drinking water at lunch | March 2013-June 2013, up to 4 months
Change in proportion of students with sugar-sweetened beverages at lunch | March 2013-June 2013, up to 4 months

REFERENCES:
- [Derived] Kenney EL, Gortmaker SL, Carter JE, Howe MC, Reiner JF, Cradock AL. Grab a Cup, Fill It Up! An Intervention to Promote the Convenience of Drinking Water and Increase Student Water Consumption During School Lunch. Am J Public Health. 2015 Sep;105(9):1777-83. doi: 10.2105/AJPH.2015.302645. Epub 2015 Jul 16. PMID 26180950